CLINICAL TRIAL: NCT01253486
Title: Use of Expressive Writing in the Cardiac Rehabilitation of Obese In-patients With Ischemic Heart Disease (IHD)
Brief Title: Expressive Writing for Heart Healing
Acronym: WrittenHeart
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Auxologico Italiano (Other)
Responsible Party: Principal Investigator, Gianluca Castelnuovo, Professor, Istituto Auxologico Italiano
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GMM 2010
Record Dates: First submitted 2010-12-02; First posted 2010-12-03 (Estimated); Last update posted 2021-02-12 (Actual); Status verified 2021-02

CONDITIONS: Ischemic Heart Disease; Obesity
Keywords: expressive writing; cardiac rehabilitation
MeSH Terms: conditions — Myocardial Ischemia; Obesity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Disease-related expressive writing (Experimental): Participants in the disease-related expressive writing condition write about their feelings about cardiac disease four times, for at least 20 minutes each time, during a two week period
  Interventions: Behavioral: Disease-related Expressive writing
- Traditional expressive writing (Active Comparator): Participants in the traditional expressive writing condition write about their feelings about one or more stressful experiences they lived in the past, for at least 20 minutes each time, during a two week period
  Interventions: Behavioral: Active Comparator: Traditional expressive writing
- Neutral writing (Sham Comparator): Participants in the neutral writing condition write about the facts about cardiac disease, for at least 20 minutes each time, during a two week period
  Interventions: Behavioral: Sham Comparator: Neutral writing
- Control condition (No Intervention): Participants in the control condition do not receive any intervention and complete only the assessments

INTERVENTIONS:
Behavioral: Disease-related Expressive writing — Participants in the disease-related expressive writing condition write about their feelings about cardiac disease four times, for at least 20 minutes each time, during a two week period.
  Arms: Disease-related expressive writing
Behavioral: Active Comparator: Traditional expressive writing — Participants in the traditional expressive writing condition write about their feelings about one or more stressful experiences they lived in the past, for at least 20 minutes each time, during a two week period
  Arms: Traditional expressive writing
Behavioral: Sham Comparator: Neutral writing — Participants in the neutral writing condition write about the facts about cardiac disease, for at least 20 minutes each time, during a two week period
  Arms: Neutral writing

SUMMARY:
This study will determine whether the psychological and physical benefits of expressive writing extend to obese in-patients with Ischemic Heart Disease (IHD)referred to cardiac rehabilitation

DETAILED DESCRIPTION:
Expressive writing, for as little as 3-5 sessions of 20 minutes, has been found to improve both physical and psychological health based on health outcome measures such as number of doctor's visits and hospital days, blood pressure control, lung and immune function, pain, anxiety and depression. Given its simplicity and obvious advantages in terms of cost-effectiveness, expressive writing has great potential as a therapeutic tool or as a means of self-help, either alone or as an adjunct to traditional therapies. This modality has not been studied in obese patients with Ischemic Heart Disease.

ELIGIBILITY:
Inclusion Criteria:

* obesity
* Ischemic Heart disease
* Signed informed consent

Exclusion Criteria:

* Visual or manual limitations that preclude reading and writing
* Unwilling to participate

Max Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2010-01; Primary Completion 2012-09 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
SF12 | 1 year
  The SF12 is a generic measure of both physical and emotional components of health-related quality of life
BDI-II | 1 year
  The Beck Depression Inventory is a measure of depressive symptoms
BDI | 1 year
  The Beck Anxiety Inventory is a measure of cognitive and somatic symptoms of anxiety
Brief-PTGI | 1 year
  The Brief Post-Traumatic Growth Inventory is a measure of positive growth following adversity

SECONDARY OUTCOMES:
BMI | 1 year
  Body Mass Index (BMI) is a measure of obesity and is calculated as weight in kilograms divided by height in meters squared
Multiple Coronary Risk Factors | 1 year
  Hypertension, HDL, LDL,
METs | 1 year
  Metabolic equivalents are a measure of exercise capacity. 1 MET represents the amount of oxygen consumed at rest and is equal to approximately 3.5 ml O2 kg-1 min-1

CONTACTS AND LOCATIONS:
Overall Officials: Gianluca Castelnuovo, Ph.D., Principal Investigator — Istituto Auxologico Italiano
Locations (1):
- San Giuseppe Hospital, Istituto Auxologico Italiano IRCSS, Verbania, Italy

REFERENCES:
- [Background] Frattaroli J. Experimental disclosure and its moderators: a meta-analysis. Psychol Bull. 2006 Nov;132(6):823-65. doi: 10.1037/0033-2909.132.6.823. PMID 17073523
- [Derived] Manzoni GM, Castelnuovo G, Molinari E. The WRITTEN-HEART study (expressive writing for heart healing): rationale and design of a randomized controlled clinical trial of expressive writing in coronary patients referred to residential cardiac rehabilitation. Health Qual Life Outcomes. 2011 Jul 8;9:51. doi: 10.1186/1477-7525-9-51. PMID 21740564
- See also: Related Info — http://www.auxologico.it